CLINICAL TRIAL: NCT03894722
Title: Effects of Polyvinylpyrrolidone Iodine Concentrations on Postoperative Trismus and Swelling Using as an Irrigation Solution During Impacted Third Molar Surgery : a Randomized Clinical Study
Brief Title: Effects of Polyvinylpyrrolidone Iodine on Postoperative Trismus and Swelling During Impacted Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cansu Gül Koca (Other)
Responsible Party: Sponsor-Investigator, Cansu Gül Koca, Head Of Department, Assistant Professor Doctor, Uşak University
Organization: Uşak University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHR: 2016-8/11
Record Dates: First submitted 2019-03-24; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Impacted Third Molar Tooth
Keywords: third molar surgery; povidone iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Device: No

ARMS (4):
- Group I (control; saline only) (Placebo Comparator): Control Group: Intraoperative irrigation with saline solution only.
  Interventions: Procedure: Control
- Group II (0.5% concentration of PVP-I ) (Experimental): Experimental Group: Intraoperative irrigation with 0.5% concentration of PVP-I solution.
  Interventions: Procedure: 0.5% concentration of PVP-I
- Group III (1% concentration of PVP-I) (Experimental): Experimental Group: Intraoperative irrigation with 1% concentration of PVP-I solution.
  Interventions: Procedure: 1 % concentration of PVP-I
- Group IV (3% concentration of PVP-I) (Experimental): Experimental Group: Intraoperative irrigation with 3% concentration of PVP-I solution.
  Interventions: Procedure: 3 % concentration of PVP-I

INTERVENTIONS:
Procedure: Control — During the third molar extraction the saline solution will be used in the control group.
  Arms: Group I (control; saline only)
Procedure: 0.5% concentration of PVP-I — During the third molar extraction 0.5% concentration of PVP-I solution will be used in the test group.
  Arms: Group II (0.5% concentration of PVP-I )
Procedure: 1 % concentration of PVP-I — During the third molar extraction 1 % concentration of PVP-I solution will be used in the test group.
  Arms: Group III (1% concentration of PVP-I)
Procedure: 3 % concentration of PVP-I — During the third molar extraction 3 % concentration of PVP-I solution will be used in the test group.
  Arms: Group IV (3% concentration of PVP-I)

SUMMARY:
The aim of the present study was to evaluate the effects of different concentrations of povidone iodine (PVP-I) on postoperative swelling and trismus when used as a coolant and irrigation solution during the surgical removal of impacted mandibular third molars.

ELIGIBILITY:
Inclusion Criteria:

* Totally impacted mandibular third molars of class C, 1, 2, and 3 according to the Pell-Gregory classification;
* Has no systemic disease

Exclusion Criteria:

* The use of medications that could interfere with the healing process;
* Smoking;
* Pregnancy or lactation;
* Presence of any condition, such as inflammation, periodontitis, gingivitis and dental abscess in the area of the impacted teeth;
* Undergoing antibiotic or anti-inflammatory drugs therapies in the 7 days before surgery;
* History of hypersensitivity to iodine;
* Has any thyroid diseases.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Postoperative Facial Swelling (assessed 3 facial lines (in millimeters) for determination of difference in facial contours before and after surgery) | Preoperative (on the day of surgery)- postoperative 2nd day-postoperative 7th day
  For the assessment of facial swelling, three facial lines (in milimeters) were measured with a digital tape on the operated side using following (4) landmarks: the external canthus of the eye, the gonion angle, the lower border of the tragus, soft pogonion and the mouth commissure
  Facial Lines between:
  1. the external canthus of the eye- the gonion angle
  2. the lower border of the tragus-the mouth commissure
  3. the lower border of the tragus- soft pogonion
Postoperative Trismus (difference in interincisal distance at the maximal mouth opening (in millimeters) before and after surgery) | Preoperative (on the day of surgery)- postoperative 2nd day-postoperative 7th day.
  The degree of trismus was assessed by measuring the distance between upper and lower incisal borders of the central incisors with a digital caliper.

REFERENCES:
- [Derived] Yuce E, Dereci O, Altin N, Koca CE, Yazan M. Effects of different polyvinylpyrrolidone iodine concentrations on trismus and swelling following third molar surgery. J Pak Med Assoc. 2020 Dec;70(12(B)):2304-2309. doi: 10.5455/JPMA.130. PMID 33475533